CLINICAL TRIAL: NCT03441412
Title: Low Dose EPInephrine to Improve Platelet Reactivity in TICagrelor-treated Subjects: A Proof of Concept Study in Healthy Volunteers (EPITIC)
Brief Title: A Study of the Effect of Epinephrine on Platelet Reactivity in Subjects Treated With Ticagrelor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Gothia Forum - Center for Clinical Trial (Other); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EudraCT 2017-003111-18
Record Dates: First submitted 2018-02-05; First posted 2018-02-22 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ticagrelor; Epinephrine; Metoprolol

STUDY DESIGN:
Intervention Model Description: The study is an experimental observational study in ten healthy volunteers. Volunteers fulfilling all of the inclusion and none of the exclusion criteria will be included. Enrollment will be continued until the required sample size is achieved (10 subjects).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ticagrelor/Epinephrine/Metoprolol (Experimental): 2 x 90 mg of ticagrelor will be administered orally to the subjects. Two hours after administration, the registrations and blood sampling are repeated after which an infusion of epinephrine diluted in glucose solution (5%) is started at a weight-adjusted rate of 0.01, 0.05, 0.10 and 0.15 μg kg-1 min-1. Each infusion will be maintained for 15 minutes.
  After the measurement at the highest dose of epinephrine, 5 mg metoprolol (Abcur, Haelsingborg , Sweden) will be given intravenously to the study subject and thereafter registrations and blood sampling will be repeated.
  Interventions: Drug: Ticagrelor 90mg; Drug: Epinephrine; Drug: Metoprolol

INTERVENTIONS:
Drug: Ticagrelor 90mg — 2 x 90 mg of ticagrelor will be administered orally to the subjects. Two hours after administration, the registrations and blood sampling are repeated after which an infusion of epinephrine diluted in glucose solution (5%) is started at a weight-adjusted rate of 0.01, 0.05, 0.10 and 0.15 μg kg-1 min-1. Each infusion will be maintained for 15 minutes.
  After the measurement at the highest dose of epinephrine, 5 mg metoprolol (Abcur, Haelsingborg , Sweden) will be given intravenously to the study subject and thereafter registrations and blood sampling will be repeated.
Drug: Epinephrine — 2 x 90 mg of ticagrelor will be administered orally to the subjects. Two hours after administration, the registrations and blood sampling are repeated after which an infusion of epinephrine diluted in glucose solution (5%) is started at a weight-adjusted rate of 0.01, 0.05, 0.10 and 0.15 μg kg-1 min-1. Each infusion will be maintained for 15 minutes.
  After the measurement at the highest dose of epinephrine, 5 mg metoprolol (Abcur, Haelsingborg , Sweden) will be given intravenously to the study subject and thereafter registrations and blood sampling will be repeated.
Drug: Metoprolol — 2 x 90 mg of ticagrelor will be administered orally to the subjects. Two hours after administration, the registrations and blood sampling are repeated after which an infusion of epinephrine diluted in glucose solution (5%) is started at a weight-adjusted rate of 0.01, 0.05, 0.10 and 0.15 μg kg-1 min-1. Each infusion will be maintained for 15 minutes.
  After the measurement at the highest dose of epinephrine, 5 mg metoprolol (Abcur, Haelsingborg , Sweden) will be given intravenously to the study subject and thereafter registrations and blood sampling will be repeated.

SUMMARY:
The study is an experimental observational study in ten healthy volunteers. Based on an in vitro study, it is hypothesize that a low dose epinephrine infusion will improve platelet function in healthy volunteers who have received ticagrelor. Volunteers fulfilling all of the inclusion and none of the exclusion criteria will be included. Enrollment will be continued until the required sample size is achieved (10 subjects).

Once informed consent is obtained, screening data will be collected to determine each subject's eligibility for study participation. The total expected duration of subject participation is 18 days, from screening visit to end of follow-up. The active participation is 8h (study procedure 4 hours, observation period 4 hours).

DETAILED DESCRIPTION:
The study is an experimental observational study in ten healthy volunteers. Volunteers fulfilling all of the inclusion and none of the exclusion criteria will be included. Enrollment will be continued until the required sample size is achieved (10 subjects).

The total expected duration of subject participation is 18 days, from screening visit to end of follow-up. The active participation is 8h (study procedure 4 hours, observation period 4 hours).

The study will include four visits in total, beginning with the written informed consent at the screening visit, followed by the study visit. A phone follow-up visit is conducted the day after the treatment and after 72h to ensure subject's well-being/ inquire if the subject have had any Adverse Event (AE).

On the treatment day, an arterial catheter for continuous invasive blood pressure registration and blood sample collection will be inserted in the radial artery. In addition, a catheter for drug administration will be inserted in the brachial vein. After baseline registration (blood pressure and pulse), blood sampling and assessment of dyspnea (Borg-scale), ticagrelor is administered orally to the subjects. Two hours after administration, the registrations and blood sampling (outcome samples) are repeated after which an infusion of epinephrine is started at a weight-adjusted rate of 0.01, 0.05, 0.10 and 0.15 μg kg-1 min-1. Each infusion will be maintained for 15 minutes. At the end of each infusion period, registrations and blood sampling are repeated. The blood pressure may increase as a result of epinephrine infusion and metoprolol will therefore be administered to investigate if it affects platelet function. Hence, after the last measurement with the highest dose of epinephrine, 5 mg metoprolol (Abcur, Haelsingborg , Sweden) will be given intravenously and thereafter registrations and blood sampling will be repeated. The infusion is then stopped and the healthy volunteers are observed for 4 hours.

All study subjects will be contacted the day after treatment and three days after treatment and asked about their wellbeing/ if they have had any AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent,
2. Males of age 18-40 years

Exclusion Criteria:

1. Any chronic physical or mental disease or disorder
2. Chronic medication of any kind
3. Any occasional doses of the following substances at least one week before the investigation due to potential interactions with ticagrelor: ketoconazole, clarithromycin, nefazodone, ritonavir, atazanavir, rifampicin, fenitoin, carbamazepin, pentobarbital , cyclosporine, verapamil, diltiazem, kinidin, heparin, enoxaparin, acetylsalicylic acid, desmopressin, digoxin, beta-blockers (e.g. metoprolol, atenolol , bisoprolol) and selective serotonin reuptake inhibitors (SSRI) (e.g. paroxetine, sertraline, citalopram). In addition non-steroidal anti-inflammatory drugs (NSAIDS) should be avoided due to an increased risk of bleeding.
4. Any occasional doses of the following substances at least one week before the investigation due to potential interactions with adrenalin: Beta-blockers ((e.g. metoprolol, atenolol , bisoprolol), tricyclic antidepressants (e.g protriptyline, maprotilin), digoxin and kinidin.
5. Any occasional doses of the following substances at least one week before the investigation due to potential interactions with metoprolol: Calcium-antagonists (verapamil, diltiazem, nifedipine), anti-arrythmics (e.g disopyramide), insulin, tricyclic antidepressants (e.g protriptyline, maprotilin), barbiturates; fentiazins and nitroglycerine.
6. Non-willingness to refrain from caffeine intake or nicotine use within 24 hours before start of treatment
7. Simultaneous participation in any other clinical study
8. Known drug abuse of any kind, or other condition that may render the subject more likely to be non-compliant to the protocol, as judged by the investigator
9. Known intolerance or contraindication to ticagrelor, adrenaline or metoprolol
10. Any disorder that may interfere with drug absorption
11. Previous intracranial bleeding
12. Any condition that in the opinion of the investigator may interfere with adherence to trial protocol

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Platelet aggregability, Area under the aggregation curve (AUC) for adenosine diphosphate (ADP)-induced platelet aggregation | The primary outcome measure will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  Area under the aggregation curve (AUC) for adenosine diphosphate (ADP)-induced platelet aggregation

SECONDARY OUTCOMES:
Platelet aggregability, Area under the aggregation curve (AUC) for arachidonic acid-aggregation. | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  Area under the aggregation curve (AUC) for arachidonic acid-aggregation.
Platelet aggregability, AUC for thrombin receptor activating peptide (TRAP)-induced aggregation. | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  AUC for thrombin receptor activating peptide (TRAP)-induced aggregation.
Platelet activation, Median fluorescence of platelets expressing PAC-1 (name of an antibody), unstimulated | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  Median fluorescence of platelets expressing PAC-1 (name of an antibody), unstimulated
Platelet activation, Percentage of platelets expressing PAC-1, unstimulated | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  Percentage of platelets expressing PAC-1, unstimulated
Platelet activation, Median fluorescence of platelets expressing PAC-1, ADP-induced | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  Median fluorescence of platelets expressing PAC-1, ADP-induced
Platelet activation, ADP-induced percentage of platelets expressing PAC-1, ADP-induced | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  ADP-induced percentage of platelets expressing PAC-1, ADP-induced
Platelet activation, Median fluorescence of platelets expressing P-selectin, unstimulated | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  Median fluorescence of platelets expressing P-selectin, unstimulated
Platelet activation, Percentage of platelets expressing P-selectin, unstimulated | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  Percentage of platelets expressing P-selectin, unstimulated
Platelet activation, Median fluorescence of platelets expressing P-selectin, ADP-induced | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  Median fluorescence of platelets expressing P-selectin, ADP-induced
Platelet activation, Percentage of platelets expressing P-selectin, ADP-induced | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  Percentage of platelets expressing P-selectin, ADP-induced
Coagulation parameters, EXTEM (name of a thromboelastometric test) Clotting time | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  EXTEM (name of a thromboelastometric test) Clotting time
Coagulation parameters, EXTEM clot formation time | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  EXTEM clot formation time
Coagulation parameters, EXTEM maximum clot firmness | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  EXTEM maximum clot firmness
Coagulation parameters, EXTEM maximum clot elasticity | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  EXTEM maximum clot elasticity
Coagulation parameters, FIBTEM (name of a thromboelastometric test) Maximum clot firmness | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  FIBTEM (name of a thromboelastometric test) Maximum clot firmness
Coagulation parameters, FIBTEM maximum clot elasticity. | The secondary outcome measures will be assessed at 7 time-points during 4 hours: before ticagrelor, 2 hours after ticagrelor, after each epinephrine infusion and after metoprolol injection.
  FIBTEM maximum clot elasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jeppsson, MD,PhD,Prof, Principal Investigator — Dep of Cardiothoracic Surgery,Sahlgrenska University Hospital,413 45 Gothenburg, Sweden
Locations (1):
- gothia Forum CTC, Gothenburg, Sweden

REFERENCES:
- [Derived] Singh S, Damen T, Nygren A, Shams Hakimi C, Ramstrom S, Dellborg M, Lindahl TL, Hesse C, Jeppsson A. Adrenaline Improves Platelet Reactivity in Ticagrelor-Treated Healthy Volunteers. Thromb Haemost. 2019 May;119(5):735-743. doi: 10.1055/s-0039-1683461. Epub 2019 Feb 19. PMID 30780166